CLINICAL TRIAL: NCT01818804
Title: The Effect of n-3 Polyunsaturated Fatty Acids on Risk Markers for Cardiovascular Disease and Inflammation in Patients With Psoriatic Arthritis
Brief Title: The Effect of n-3 Polyunsaturated Fatty Acids in Patients With Psoriatic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Salome Kristensen, MD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-20120076
Record Dates: First submitted 2013-03-20; First posted 2013-03-27 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- n-3PUFA (Active Comparator): n-3 polyunsaturated fattyacids from fish oil
  Interventions: Dietary Supplement: n-3PUFA
- olive oil (Placebo Comparator): Olive oil
  Interventions: Dietary Supplement: olive oil

INTERVENTIONS:
Dietary Supplement: n-3PUFA
  Other Names: n-3 polyunsaturated fattyacids from fishoil
  Arms: n-3PUFA
Dietary Supplement: olive oil
  Arms: olive oil

SUMMARY:
Background: There is evidence for a high cardiovascular risk in rheumatic and inflammatory diseases . Recent evidence suggest that psoriatic arthritis is also associated with an increased cardiovascular risk with accelerated atherosclerosis and increased cardiovascular risk. However, data regarding cardiovascular comorbidity and cardiovascular risk factors in patients with psoriatic arthritis are limited.

Objective: The aim of this study is to investigate the effect of daily supplementation with 3 g n-3 polyunsaturated fatty acids on risk markers for cardiovascular disease and inflammation in patients with psoriatic arthritis.

Design: Randomized double-blind, placebo-controlled, multicenter trial with n-3 polyunsaturated fatty acids in patient with psoriatic arthritis.

Setting: Departments of Rheumatology, Nephrology and Cardiology at Aalborg University Hospital and Vendsyssel Hospital in Region Northern Denmark

Participants: 156 men and women aged > 18 years with psoriatic arthritis classified by the CASPAR criteria will be included. Exclusion criteria: cardiac arrhythmias, conduction disturbances, treatment with biological drugs or oral corticosteroids. Inclusion time: spring 2013 to spring 2015.

Method: The following data will be collected for each participant: Interview including dietary records, assessment of tender and swollen joints, enthesitis, dactylitis, patient global assessment of disease activity (Visual Analogue Scale ), global assessment of pain (Visual Analogue Scale), psoriatic skin involvement by Psoriatic Area and Severity Index (PASI), laboratory parameters of disease activity and risk markers of cardiovascular disease.

For detection of early cardiovascular risk markers Heart Rate Variability (HRV) and Pulse Wave Velocity (PWV) will be performed.

Main outcome measures: The primary endpoint will be HRV and secondary endpoints will be PWV, inflammatory activity and use of analgesics.

The trial is approved by The local Ethics Committee, registration number N20120076

DETAILED DESCRIPTION:
Method Study design: The study was designed as a randomized, double-blind, placebo-controlled, multicenter trial. The patients were randomly assigned in blocks of five by a computer-generated block sequence. For 24 weeks patients were assigned to daily intake of 6 capsules containing either 3 g of n-3 PUFA (50% EPA and 50% DHA) from fish oil capsules or 3 g of olive oil (approximately 80% of oleic acid and 20% linoleic acid). All the investigators, patients and research staff were blinded to the supplementation codes. Patients were asked to maintain their usual diet during the whole study. The study was conducted in accordance with the Declaration of Helsinki and Good clinical practice (GCP).

Subjects: Patients with PsA defined by Classification criteria for psoriatic arthritis (CASPAR) (25) were enrolled from the Departments of Rheumatology, Aalborg University Hospital and Department of Rheumatology, Vendsyssel Hospital, in Denmark. The inclusion criteria were PsA in adult above 18 years of age with any disease activity while exclusion criteria were documented cardiac arrhythmias, treatment with biological drugs or treatment with oral corticosteroids.

Compliance was assessed by counting capsules during the last visit. Patients were defined as non-compliant if >150 capsules were returned and those were not included in the per-protocol analysis.

All participants gave their written informed consent and the regional ethics committee of Northern Region Denmark, approved the study.

Clinical assessment: Patients were assessed at baseline, after 12 weeks of supplement and after 24 weeks. At baseline, duration of disease, medical history, smoking habits and diet were obtained Medical history of diabetes mellitus, hypertension and dyslipidemia were assessed and was defined as present if the patient received dietary or medical therapy for the condition. A food questionnaire was used to assess patients' fish consumption at lunch and dinner. A score for fish intake was given according to the following: never eat fish = 1; eat fish once a month =2; eat fish two to three times a month = 3; eat fish once a week = 4; eat fish two to three times a week = 5; and eat fish at least once daily = 6.

At each visit conventional cardiovascular risk factors such as smoking habits, blood pressure, body mass index (BMI) and waist to hip ratio (WHR) were assessed in all patients. Additionally, a clinical evaluation was performed, consisting of 68 tender joint count, 66 swollen joint count, disease activity score (DAS) and psoriatic skin area involvement (PASI).

Blood samples: Blood samples were taken non-fasting in the morning for assessment of fatty acid composition of granulocytes and routine laboratory evaluation. Granulocytes were isolated from whole blood, and lipids were extracted and fatty acids esterified as previously reported (26). The fatty acid composition in granulocytes were determined by gas chromatography with a Chrompack CP-9002 gas chromatograph (Varian, Middelberg, The Netherlands) and expressed as weight percent (wt. %) of total fatty acids.

HRV: Five min HRV recordings were obtained with SphygmoCor Technology (SphygmoCor, Software version 8.2; AtCor Medical, Sydney, NSW, Australia).

HRV was recorded in each patient according to current recommendations (27). The measurements were obtained in the morning hours after resting for 15 min in a room with a constant temperature of 20°C. Patients were instructed not to smoke and avoid alcohol and caffeine-containing beverages within 12 h prior to investigation. A trained technician blinded to the type of supplement performed these analyses. The patients were placed in a supine position (resting) for 10 min, breathing spontaneously without talking. HRV were analysed in the time-domain and the following variables were used:

* RR: mean of all normal RR intervals during the 5 min recording
* SDNN: standard deviation of all normal RR intervals in the 5 min recording
* SDNNindex: mean of the standard deviation of all the normal RR intervals.
* pNN50: percentage of successive RR-interval differences > 50 ms
* RMSSD: square root of the mean of the sum of the squares of differences between adjacent intervals

PWV: PWV and pulse wave analysis were performed non-invasively with the Sphygmocor system (AtCor Medical, Sydney, NSW, Australia), as described previously (28) and according to international recommendations (29). All measurements were made in duplicate by a single trained operator and the mean of the two values was used in the analysis.

Carotid-radial and carotid-femoral PVW was measured using arterial tonometry. All measurements were performed on the right side extremities. The surface distance was measured with a tape measure as a straight line from the suprasternal notch to the carotid location (proximal pulse) and subtracted the distance from the suprasternal notch to the radial or femoral location (distal pulse) (30,31). The pressure wave transit time was determined as the time between the R-wave of the ECG and the proximal pulse subtracted from the time between the R-wave of the ECG and the distal pulse. PWV was subsequently calculated by dividing the surface distance by the pressure wave transit time.

The central BP was estimated using the SphygmoCor® device. After 10 min of rest in the supine position, brachial BP was measured three times at 2-min intervals on the left arm with the automatic Microlife® device, and the last measurement was taken as representative of brachial artery BP. Hereafter, radial artery pressure waveforms of the right arm were sampled. Using the validated generalized transfer function, central BP was estimated using brachial systolic and diastolic BP (32,33). Aortic augmentation index (AIx) was standardized to a heart rate of 75 beat per minute to minimize the effect of the heart rate. Only measurements with T1 (the time to the initial upstroke of the pressure wave) >80 and <150 ms and augmentation index (AI, the difference between the first and second peak of the arterial waveform as percentage of the pulse pressure) <50% and operator index (an arbitrary number between 1 and 100 describing the quality of the derived pulse wave) >80 were accepted according to recommendations (AtCor Medical® website).

Statistical Analysis All statistical analyses were performed using STATA version13 (StataCorp LP, TX, US) We hypothesized that intervention with n-3 PUFA would increase the HRV parameter RR by 0.5 of a standard deviation (SD).

To achieve this at p<0.05 and 1-β = 0.80 we needed a sample size with 63 subjects in each group.

The difference in the continuous outcomes between baseline and 24 weeks after randomization was compared between the two treatment groups in a one-sided analysis of variance (ANOVA). Equality of variances between the treatment groups was assessed using Bartlett's test. Due to the potential for confounding after the random treatment assignment an analysis of covariance (ANCOVA) was performed. Prior to this analysis a check for collinearity between the covariates was performed and the model was modified accordingly. In this model equality of variances was assessed using Levene's test.

The total number of parameters in the models was restricted to one tenth of the number of study participants or number of each category when specifying the models.

All analyses were performed both as intention to treat (none of the patients are excluded and the patients are analyzed according to the randomization scheme) and per-protocol (patients who complete the entire clinical trial according to the protocol) analyses. The analyses were controlled for age, sex, smoking status, presence and absence of diabetes mellitus, hypertension and hypercholesterolemia, the use of nonsteroidal anti-inflammatory drugs (NSAID) and disease activity scores.

Differences were considered significant with a p-value of <0.05 (two-tailed).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged > 18 years with
* Psoriatic arthritis classified by the CASPAR criteria
* written informed consent

Exclusion Criteria:

* Treatment with biological drugs
* Treatment with oral corticosteroids
* cardiac arrhythmias

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salome Kristensen, MD, Principal Investigator — Aalborg Universityhospital, Department og Rheumatology; Jeppe H Christensen, Professor, Study Director — Aalborg University Hospital, Department of Nephrology
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, Department of Rheumatology, Aalborg
  - Vendsyssel Hospital in Region Northern Denmark, Department of Rheumatology, Hjørring

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Holm Nielsen S, Sardar S, Siebuhr AS, Schlemmer A, Schmidt EB, Bay-Jensen AC, Karsdal MA, Christensen JH, Kristensen S. Effect of n-3 PUFA on extracellular matrix protein turnover in patients with psoriatic arthritis: a randomized, double-blind, placebo-controlled trial. Rheumatol Int. 2021 Jun;41(6):1065-1077. doi: 10.1007/s00296-021-04861-z. Epub 2021 Apr 22. PMID 33885930
- [Derived] Kristensen S, Schmidt EB, Schlemmer A, Rasmussen C, Lindgreen E, Johansen MB, Christensen JH. The effect of marine n-3 polyunsaturated fatty acids on cardiac autonomic and hemodynamic function in patients with psoriatic arthritis: a randomised, double-blind, placebo-controlled trial. Lipids Health Dis. 2016 Dec 12;15(1):216. doi: 10.1186/s12944-016-0382-5. PMID 27955663

RESULTS

PARTICIPANT FLOW:
Groups:
- n-3PUFA: n-3 polyunsaturated fattyacids from fish oil
  3 g of n-3PUFA pr day
- Olive Oil: Olive oil
  3 g of olive oil pr day
Period: Overall Study
Arm/Group | n-3PUFA | Olive Oil
Started | 73 | 72
Completed | 68 | 65
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- n-3PUFA: n-3 polyunsaturated fattyacids from fish oil
  n-3PUFA
- Total: Total of all reporting groups
Arm/Group | n-3PUFA | Olive Oil | Total
Number analyzed (Participants) | 73 | 72 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 62 | 126
  >=65 years | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (11.4) | 50.7 (11.5) | 52 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 83
  Male | 33 | 29 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 73 | 72 | 145
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 73 | 72 | 145

OUTCOME MEASURES:

1. Primary Outcome: Change in Heart Rate Variability (HRV) Measure
Description: Heart Rate variability, non-invasive measurement for the autonom regulation of the heart associated with risk of cardiovascular disease
Time Frame: 24 week
Measure: Mean (95% Confidence Interval); unit: ms
Arm/Group | n-3PUFA | Olive Oil
Number analyzed (Participants) | 68 | 60
ms | 13.38 [-5.06 to 31.83] | -13.48 [-35 to -8.69]

2. Secondary Outcome: Change in PWV
Description: Pulse wave Velocity, non-invasive measurement for arterioscleroses
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: m/s
Arm/Group | n-3PUFA | Olive Oil
Number analyzed (Participants) | 68 | 60
m/s | 0.01 [-0.44 to 0.46] | 0.08 [-0.33 to 0.49]

3. Other Pre Specified Outcome: Change in Disease Activity
Description: Disease activity score (DAS-28) is a system developed and validated by the EULAR (European League Against Rheumatism) to measure the progress and improvement of Rheumatoid Arthritis. DAS28 is often used in clinical trials for arthritis
  DAS28 values range from 2.0 to 10.0 while higher values mean a higher disease activity. A DAS 28 below the value of 2.6 is interpreted as Remission.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | n-3PUFA | Olive Oil
Number analyzed (Participants) | 63 | 67
units on a scale | -0.22 [-0.38 to -0.05] | -0.05 [-0.25 to 0.15]

ADVERSE EVENTS:
Arm/Group | n-3PUFA | Olive Oil
Serious Adverse Events (participants affected / at risk) | 1/73 | 3/72
Other Adverse Events (participants affected / at risk) | 0/73 | 2/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | n-3PUFA (N=73) | Olive Oil (N=72)
Infection (Infections and infestations) | 1 (1) | 0 (0) — Wound on a finger became infected and the patient was addmited to the hospital for treatment with antibiotics
Joint inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — The patient had a major flare in arthritis and was addmitted to the hospital for treatment
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) — The patient was addmitted to the hospital because of sudden dissiness. The results showed benign vertigo
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | n-3PUFA (N=73) | Olive Oil (N=72)
nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes